CLINICAL TRIAL: NCT01801644
Title: Neoadjuvant Gemcitabine and Cisplatin in Locally Advanced Bladder Cancer
Brief Title: Neoadjuvant Chemotherapy in Locally Advanced Bladder Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barmherzige Brüder Vienna (Other)
Responsible Party: Principal Investigator, Johannes Meran, Prof. Dr.Johannes Meran, Barmherzige Brüder Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bladder Cancer-001; Bladder Cancer-001 (Other: Barmherzige Brüder, Austria)
Record Dates: First submitted 2013-02-15; First posted 2013-03-01 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; neoadjuvant chemotherapy; gem/cis
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gemcitabine plus cisplatin (Experimental): gemcitabine plus cisplatin: 3 cycles of gemcitabine 1000 mg/m2 on days 1,8,15 as a 30 minute infusion and cisplatin 70 mg/m2 on day 1 as an 2 hour infusion will be applied
  Interventions: Drug: gemcitabine plus cisplatin

INTERVENTIONS:
Drug: gemcitabine plus cisplatin — gemcitabine 1000 mg/m2 on days 1,8,15 as a 30 minute infusion followed by cisplatin 70 mg/m2 on day 1 as an 2 hour infusion
  Other Names: gemzar (gemcitabine) plus cisplatin (= cisplatin)

SUMMARY:
To evaluate the efficacy and safety of neoadjuvant gemcitabine and cisplatin (gem/cis) in locally advanced bladder cancer.

DETAILED DESCRIPTION:
Patients with locally advanced transitional cell bladder cancer receive 3 cycles of neoadjuvant gemcitabine/cisplatin before radical cystectomy.

Patients with histologically confirmed clinical stage T2-T4a, N0-2 bladder cancer are going to be included. After CT scan of the thorax and abdomen plus MRI of the pelvis patient receive chemotherapy.

Pathologic response rate will be assessed after surgery by the institutional pathologic review. Safety is going to be assessed according to the National Cancer Institute Common Toxicity Criteria (CTC,version 3.0).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* histologically confirmed stage T2, T3 or T4a urothelial bladder cancer with N0-N2
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* bone marrow reserve (neutrophil count >1500 cells per μL,platelet count >100 000 per μL) count
* hepatic function (serum bilirubin <2,5 times the upper limit of normal, serum aminotransferase ≤2,5 times the upper limit of normal).
* renal function with a creatinine clearance >60ml/min

Exclusion Criteria:

* metastatic disease
* serious or uncontrolled concurrent medical illness
* pregnancy
* history of other malignancies (with the exception of excised cervical or basal skin or squamous-cell carcinoma)
* non-transitional cell bladder cancer
* creatinine clearance <60ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-04; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
pathologic response rate | at time of surgery
  evaluation of the pathologic response rate after 3 cycles of neoadjuvant gemcitabine/cisplatin at time of radical cystectomy

SECONDARY OUTCOMES:
safety, number of participants with adverse events and grade of adverse events | adverse events will be evaluated after every 6 months
  to assess the safety of neoadjuvant gemcitabine/cisplatin in bladder cancer

OTHER OUTCOMES:
progression free survival (PFS) | up to 5 years after including the last patient
  pfs will be assessed avery 3 months in the first year after radical cystectomy, every 6 months in the second year, and yearly from the 3rd year up to a minimum follow up of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Meran, M.D., Principal Investigator — Barmherzige Brüder Vienna
Locations (1):
- Barmherzige Brüder Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Dash A, Pettus JA 4th, Herr HW, Bochner BH, Dalbagni G, Donat SM, Russo P, Boyle MG, Milowsky MI, Bajorin DF. A role for neoadjuvant gemcitabine plus cisplatin in muscle-invasive urothelial carcinoma of the bladder: a retrospective experience. Cancer. 2008 Nov 1;113(9):2471-7. doi: 10.1002/cncr.23848. PMID 18823036
- [Result] Tolerability of neoadjuvant chemotherapy with gemcitabine plus cisplatin in elderly (older than age 65) patients (pts) with muscle-invasive urothelial cancer. D. Niedersuess-Beke, B. Gruenberger, T. Puntus, W. Bauer, M. Lamche, P. Schramek, J. G. Meran; Barmherzige Brueder Hospital, Vienna, Austria; Goettlicher Heiland Hospital, Vienna, Austria ´ J Clin Oncol 29: 2011 (suppl 7; abstr 296)